CLINICAL TRIAL: NCT05980156
Title: Clinical Trial to Evaluate Intermittent Screening and Treatment and Intermittent Preventive Treatment of Malaria in Asymptomatic Schoolchildren to Decrease P. Falciparum Infection and Transmission: Phase 2 Comparing Drug Regimens
Brief Title: Comparing Chemoprevention Drugs for School-based Malaria Control
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: Kamuzu University of Health Sciences (Other); Doris Duke Charitable Foundation (Other)
Responsible Party: Principal Investigator, Lauren Cohee, Assistant Professor of Pediatrics, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HP-00098250v3
Record Dates: First submitted 2023-07-28; First posted 2023-08-07 (Actual); Last update posted 2023-08-07 (Actual); Status verified 2023-08

CONDITIONS: Malaria,Falciparum; Anemia in Children
Keywords: malaria; school; chemoprevention; preventive treatment; education; cognitive function; adolescent; hemoglobin
MeSH Terms: conditions — Malaria, Falciparum; Malaria | interventions — Chloroquine; Hydroxychloroquine; fanasil, pyrimethamine drug combination

STUDY DESIGN:
Intervention Model Description: Students were randomized to three arms in the original trial. In this follow-on study, students will remain in their study arms. Arm 1 which previously received intermittent screening-and-treatment will now receive intermittent preventive treatment with sulfadoxine-pyrimethamine plus chloroquine. Arm 2 which received intermittent preventive treatment with dihydroartemisinin-piperaquine will again receive intermittent preventive treatment with dihydroartemisinin-piperaquine. Arm 3 the control arm will continue as a control. Females 10 years and older (potentially post-menarche) in Arms 1 and 2 will receive chloroquine alone.
Who Masked: Outcomes Assessor
Masking Description: Laboratory technicians processing samples will be blinded to participant's study arm.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intermittent Preventive Treatment with dihydroartemisinin-piperaquine (IPT-DP) (Experimental): All students are treated at each intervention. Treatment will be with DP (females less than 10 years old and all males) or chloroquine (females 10 years old or older).
  Interventions: Drug: Dihydroartemisinin-Piperaquine; Drug: Chloroquine
- Intermittent Preventive Treatment with sulfadoxine-pyrimethamine plus chloroquine (IPT-SPCQ) (Experimental): All students are treated at each intervention. Treatment will be with SP + CQ (females less than 10 years old and all males) or chloroquine (females 10 years old or older).
  Interventions: Drug: Chloroquine; Drug: Sulfadoxine pyrimethamine
- Control (No Intervention): Students will not receive preventive treatment.

INTERVENTIONS:
Drug: Dihydroartemisinin-Piperaquine — Treatment will be with DP (females less than 10 years old and all males) or chloroquine alone (females 10 years old or older).
  Other Names: DP; D-Artepp; DuoCotecxin; Artekin; Eurartesim; Ridmal
  Arms: Intermittent Preventive Treatment with dihydroartemisinin-piperaquine (IPT-DP)
Drug: Chloroquine — Treatment of females 10 years old and older in Arm 1 and treatment of all participants in Arm 2.
  Other Names: Aralen; Hydroxychloroquine; Lariago
  Arms: Intermittent Preventive Treatment with dihydroartemisinin-piperaquine (IPT-DP); Intermittent Preventive Treatment with sulfadoxine-pyrimethamine plus chloroquine (IPT-SPCQ)
Drug: Sulfadoxine pyrimethamine — Treatment will be with SP and chloroquine (females less than 10 years old and all males) or chloroquine alone (females 10 years old or older).
  Other Names: SP
  Arms: Intermittent Preventive Treatment with sulfadoxine-pyrimethamine plus chloroquine (IPT-SPCQ)

SUMMARY:
This is an individually randomized, controlled, single blind three arm clinical trial of malaria chemoprevention strategies Arm 1: Intermittent preventive treatment with dihydroartemisinin-piperaquine (IPT-DP). Arm 2: Intermittent preventive treatment with sulfadoxine-pyrimethamine (SP) plus chloroquine (CQ) (IPT-SPCQ). Arm 3: Control - students will receive standard of care (no preventive treatment). Outcomes include P. falciparum infection and parasite density, anemia, cognitive function and educational testing, as well as infection prevalence in young children sleeping student's households to assess the impact on transmission.

DETAILED DESCRIPTION:
Students attending a single primary school in Machinga District, Malawi who were enrolled in NCT05244954 were offered enrollment in this follow-on study. The intervention will be conducted every 6-weeks during the two school terms which coincide with peak malaria transmission. Students in the IPT-DP arm will be treated with with dihydroartemisinin-piperaquine (DP) (females less than 10 years old and all males) or chloroquine (females 10 years old or older. Students in the IPT-SPCQ arm will be treated with sulfadoxine-pyrimethamine plus chloroquine (females less than 10 years old and all males) or chloroquine alone (females 10 years old or older).

ELIGIBILITY:
Inclusion Criteria:

Students (enrolled in the primary intervention)

* Previously enrolled in NCT05244954
* Currently enrolled in the study school
* Plan to attend the study school for the remainder of the school year
* Parent/guardian available to provide written informed consent Younger children in participant households (enrolled in the Household Prevalence survey)
* Slept in the household for most nights in the last month
* Age 6-59 months
* Parent/guardian available to provide written informed consent

Exclusion Criteria:

Students (enrolled in the primary intervention)

* Current evidence of severe malaria or danger signs
* Known adverse reaction to the study drugs
* History of cardiac problems or fainting
* Taking medications known to prolong QT
* Family history of prolonged QT
* Taking trimethoprim-sulfamethoxazole aka Bactrim or Cotrimoxazole
* Epilepsy
* Psoriasis Household members (enrolled in the Household Prevalence survey)
* Household with more than one school-age child enrolled in the study
* Current evidence of severe malaria or danger signs

Min Age: 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 646 (Actual)
Dates: Start 2023-02-13 (Actual); Primary Completion 2023-07-28 (Actual); Study Completion 2023-07-28 (Actual)

PRIMARY OUTCOMES:
Number of participants with P. falciparum infection | 6-8 weeks after the last intervention
  detected by polymerase chain reaction (PCR, binary)

SECONDARY OUTCOMES:
Number of participants with anemia | 6-8 weeks after the last intervention
  World Health Organization age-sex definitions (binary)
Mean hemoglobin concentration | 6-8 weeks after the last intervention
  g/dL (continuous)
Total parasite density | 6-8 weeks after the last intervention
  log transformed (continuous)
Rate of clinical malaria | through study completions, approximately 6 months
  cumulative incidence
P. falciparum prevalence among children less than 5 years old living in households with study participants | 6-8 weeks after the last intervention
  detected by PCR
sustained attention | 6-8 weeks after the last intervention
  code transmission test score (continuous)
selective attention | 6-8 weeks after the last intervention
  selective attention test score (continuous)
Literacy skills | 6-8 weeks after the last intervention
  onetest reading test score (continuous)
Math skills | 6-8 weeks after the last intervention
  onetest math score (continuous)

CONTACTS AND LOCATIONS:
Overall Officials: Lauren Cohee, MD MS, Principal Investigator — University of Maryland, Baltimore
Locations (1):
- Kamuzu University of Health Sciences, Blantyre, Malawi

IPD SHARING:
Plan to Share IPD: Yes
all individual participant data that underlie results in a publication
Supporting Information: Study Protocol, ICF
Time Frame: After results publication
Access Criteria: Public access with registration to allow tracking

REFERENCES:
- [Background] Cohee LM, Valim C, Coalson JE, Nyambalo A, Chilombe M, Ngwira A, Bauleni A, Seydel KB, Wilson ML, Taylor TE, Mathanga DP, Laufer MK. School-based screening and treatment may reduce P. falciparum transmission. Sci Rep. 2021 Mar 25;11(1):6905. doi: 10.1038/s41598-021-86450-5. PMID 33767384
- [Background] Cohee LM, Opondo C, Clarke SE, Halliday KE, Cano J, Shipper AG, Barger-Kamate B, Djimde A, Diarra S, Dokras A, Kamya MR, Lutumba P, Ly AB, Nankabirwa JI, Njagi JK, Maiga H, Maiteki-Sebuguzi C, Matangila J, Okello G, Rohner F, Roschnik N, Rouhani S, Sissoko MS, Staedke SG, Thera MA, Turner EL, Van Geertruyden JP, Zimmerman MB, Jukes MCH, Brooker SJ, Allen E, Laufer MK, Chico RM. Preventive malaria treatment among school-aged children in sub-Saharan Africa: a systematic review and meta-analyses. Lancet Glob Health. 2020 Dec;8(12):e1499-e1511. doi: 10.1016/S2214-109X(20)30325-9. Epub 2020 Oct 22. PMID 33222799